CLINICAL TRIAL: NCT02647125
Title: A Phase II Study of Comparing Huachansu Combination With Thoracic Radiotherapy Versus Radiotherapy Alone For Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Comparing Huachansu Plus Thoracic RT Versus RT Alone For ESCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai3
Record Dates: First submitted 2015-12-12; First posted 2016-01-06 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — huachansu

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huachansu Arm (Experimental): Patients in this arm will receive a treatment of Huachansu combined with thoracic radiotherapy.
  Interventions: Drug: Huachansu; Radiation: thoracic radiation
- Control Arm (Active Comparator): Patients in this arm will receive thoracic radiotherapy alone.
  Interventions: Radiation: thoracic radiation

INTERVENTIONS:
Drug: Huachansu — Huachansu 20 ml/m2/d, intervenous infusion, once a day, 5 times per week, during the period of radiation.
  Arms: Huachansu Arm
Radiation: thoracic radiation — A total dose of 61.2 Gy will be delivered in 34 fractions at 1.8 Gy/fraction, 5 fractions per week in 6.8 weeks.

SUMMARY:
This primary objective of the trial is to study whether the local control of Huachansu plus thoracic radiotherapy is better compared to thoracic radiotherapy alone for patients with esophageal squamous cell carcinoma. It's a phase II study, 134 patients are expected to be recruited into the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Joined the study voluntarily and signed informed consent form.
2. Age >75 or age 18-75 who are intolerant of or reject intravenous chemotherapy.
3. Both genders.
4. Esophageal squamous cell carcinoma confirmed by pathology.
5. Local advanced esophageal squamous cell carcinoma (T2-4N0-1M0-1a,TxN1M0-1a,TxNxM1a, AJCC 6th).
6. No radiotherapy, chemotherapy or other treatments prior to enrollment.
7. PS ECOG 0-2，wight loss<30% during the latest 6 months.
8. Life expectancy of more than 3 months.
9. Hemoglobin（Hb）≥9 g/dL,WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L platelet count (Pt) ≥100x 109/L.Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL<1.5 x ULN.Renal function: creatinine < 1.5 x ULN.
10. No immuno-deficiency
11. No heart diseases that need cardiac glycoside
12. Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

1. Complete esophageal obstruction.
2. Deep esophageal ulcer.
3. Esophageal perforation.
4. Haematemesis.
5. After surgery, exploratory thoracotomy, radiotherapy, chemotherapy, or targeting therapy.
6. Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years.
7. Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives.
8. Drug addiction,Alcoholism or AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Local control rate | the date of randomization until progression inside the irradiation field, up to 3 years.
  The outcome measure will be assessed by every 3-month follow-up examinations.

SECONDARY OUTCOMES:
overall survival | the date of randomization until the death or the last follow up of the patients, up to 3 years.
  The survival time from date of randomization to the day of death or the last follow-up.
progress-free survival | the date of randomization until progression or death from any cause, up to 3 years
  Measured from date of randomization until progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Shen J, Chen Y, Zhou J, Luo H, Deng J, Ai D, Zhu H, Hao S, Zhao K. Phase II trial of radiotherapy plus Huachansu in elderly or chemotherapy-ineligible patients with locally advanced esophageal squamous cell carcinoma. Oncologist. 2025 Oct 1;30(10):oyaf325. doi: 10.1093/oncolo/oyaf325. PMID 41021440